CLINICAL TRIAL: NCT01552616
Title: Evaluation of Thermal-aided Muscle Activation in Intensive Care Unit (ICU) Patients - A PILOT Study
Brief Title: Safety and Performance of Muscle Activation for Critical Care Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment
Sponsor: Niveus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NMSA
Record Dates: First submitted 2012-02-20; First posted 2012-03-13 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Critically-ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Activation Treatment (Experimental)
  Interventions: Procedure: Thermal-aided muscle activation
- Usual Care (No Intervention): This arm will not receive any study-motivated intervention. Subjects will receive usual care, but will participate in outcomes assessments.

INTERVENTIONS:
Procedure: Thermal-aided muscle activation — Thermal-aided muscle activation therapy will be provided to patients twice daily. Treatment will begin within 24 hours of admission and continue until patients are significantly ambulatory.
  Arms: Activation Treatment

SUMMARY:
Critically-ill patients who have long stays in the hospital often face prolonged periods of bed rest. It is known that these patient develop profound weakness and debilitation. The effectiveness of existing muscle activation devices that could otherwise prevent the onset of debilitation in an immobilized patient has not been demonstrated widely in this cohort. It is hypothesized that using thermal methods to augment existing muscle activation techniques may demonstrate improved performance with no corresponding change in the safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Patient is enrolled within 60 hours of admission to the ICU
* Patient expected to be subject to bedrest in the ICU for > 96 hours

Exclusion Criteria:

* Patient is age < 18 years at time of consent
* Patient is pregnant
* Patient is moribund
* Patient has an implanted pacemaker/defibrillator
* Patient has a documented diagnosis of epilepsy
* Patient has implanted femoral rods
* Patient has leg or pelvic trauma that limits mobility
* Patient has recent trauma resulting in GCS < 5
* Patient lacks ability to walk without assistance prior to acute ICU admission
* Patient has neuromuscular disease or abnormalities
* Patient is morbidly obese (BMI > 40)
* Patient has a cognitive impairment or inability to follow commands prior to acute ICU admission
* Patient was transferred after > 48 hours at another acute care institution
* Enrollment in another investigational device or drug trial that could compromise the conduct or results of the study
* Evidence of disease or condition that, in the opinion of the physician, may compromise the conduct of or results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Muscle Activation Effectiveness | Day of ICU Discharge, expected on average 5 days
  Research team will assess whether or not visible or palpable muscle contractions can be activated in the target patient population.

SECONDARY OUTCOMES:
Muscle Mass | At enrollment, at ICU discharge (expected average days), at hospital discharge (expected average 10 days)
  Muscle mass will be measured at several time points during the patient stay.
Muscle Strength | At enrollment, at ICU discharge (expected average days), at hospital discharge (expected average 10 days)
  Muscle strength will be assessed using MRC scales at various time points throughout the study
Activities of Daily Living | At hospital discharge (expected average 10 days)
  The subject's proficiencies and independence in Activities of Daily Living will be assessed prior to hospital discharge.
Six Minute Walk | At time of first ambulation (expected average 7 days), at hospital discharge (expected average 10 days)
  A 6 minute walk test administered per ATS guidelines will be undertaken by all patients prior to discharge. When possible at least 2 six minute walk tests will be administered.
Time to ambulation | During timeframe when patient moves out of bed, expected on average 5 - 8 days into study
  The time needed for a patient who had previously been subjected to bed rest to ambulate will be noted through chart review and nursing interviews.
Length of stay | At end of study, expected on average after 10 days
  The subject's length of stay will be recorded from chart review.
Ventilator Dependency | During active ventilation and weaning period, expected to last on average 4 - 7 days per patient
  Chart review will be used to determine the number of ventilator days and the ventilator weaning time for each subject

CONTACTS AND LOCATIONS:
Overall Officials: Mark Tidswell, MD, Principal Investigator — Baystate Medical Center
Locations (5):
- United States (5):
  - University of Arizona Medical Center, Tucson, Arizona
  - Franklin Square Medical Center, Baltimore, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Ohio State University Medical Center, Columbus, Ohio